CLINICAL TRIAL: NCT03307772
Title: A Randomized, Triple-blind Placebo-controlled Single Center Trial to Evaluate the Immune Response to the Consumption of a Minidrink Containing a Combination of Lactobacillus GG and Fructooligosaccharides in Patients With Recurrent Herpes Labialis
Brief Title: Immune Response to the Consumption of Lactobacillus GG and FOS in Patients With Recurrent Herpes Labialis
Acronym: EVIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-SBUS-2-GRA-01 A
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Herpes Labialis
Keywords: lactobacillus; Herpes Labialis; immune response
MeSH Terms: conditions — Herpes Labialis | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo drink (Placebo Comparator): The placebo drink consists of fermented low-fat milk with no added Lactobacillus GG.(placebo)
  Interventions: Dietary Supplement: Placebo
- LGG Drink ( (Active Comparator): The probiotic drink consists of fermented low-fat milk with added Lactobacillus GG. (probiotics)
  Interventions: Dietary Supplement: Probiotics
- FOS Drink (Active Comparator): The prebiotics drink consists of fermented low-fat milk with fructooligosaccharides. (prebiotics)
  Interventions: Dietary Supplement: Prebiotics
- LGG e FOS Drink (Active Comparator): The probiotics and prebiotics drink consists of acidified low-fat milk with added Lactobacillus GG and fructooligosaccharides (prebiotics and probiotics)
  Interventions: Dietary Supplement: Prebiotics and Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: LGG Drink (
Dietary Supplement: Prebiotics
  Arms: FOS Drink
Dietary Supplement: Prebiotics and Probiotics
  Arms: LGG e FOS Drink
Dietary Supplement: Placebo
  Arms: placebo drink

SUMMARY:
Background: Herpes labialis is the result of the presence of Herplex Simplex Virus -1 (HSV-1) and is a common disease in the population. Because of its visibility it has a serious impact on social life and the feeling of well-being in people who suffer from this disease. Until now there is no effective treatment and no remedy for prevention of the virus outbreak.

Prebiotics and probiotics have both been shown to have a favorable and supportive effect on the immune system in different health conditions such as influenza, atopic dermatitis and diarrhea. So far no study has addressed the effect of the consumption of pre- and/or probiotics in a population with recurrent herpes labialis.

Aim of the study: The present study investigated the effect of pre- or probiotics or a combination of the two on the recurrence of herpes labialis lesions as well as on the immune system in general.

Design: 78 Patients were eligible to participate in the study and after a run-in period of two weeks consuming a placebo minidrink were randomized to one of the four experimental groups, these were: placebo minidrink (n=), prebiotic (fructooligosaccharides) minidrink (n=), probiotic (Lactobacillus rhamnosus GG or LGG) minidrink (n=) or a minidrink containing a combination of a pre- and probiotic. These minidrinks were consumed for another 5 weeks. At day 33 of the study the lip most prone to the development of a lesion was stimulated with UVB in order to provoke a lesion. During the entire study period subjects were checked for any clinical signs of a lesion, completed a self-assessment regarding the lesion and a quality of life questionnaire at baseline (day 14) and the end of the study (day 49). In addition, a blood sample was collected at baseline and at the end of the study to be analyzed for general and HSV-specific antibodies, intracellular cytokine concentrations and parameters of the innate immune response such as natural killer cell activity and phagocytosis.

DETAILED DESCRIPTION:
The present study showed that the daily consumption of a minidrink containing either only Lactobacillus rhamnosus or a combination of Lactobacillus rhamnosus and fructooligosaccharides significantly decreased both the occurrence and the incidence of Herpes labialis lesions after stimulation with UVR in a population with recurrent Herpes labialis. No difference in the function of either CD8+ T lymphocytes or natural killer cells was found, nevertheless a trend, that did not reach statistical significance, was observed for some of the immunological analyses pointing out towards an immunemodulating effect of probiotic or pre- and probiotic combination minidrink on the adaptive immune system. The end of study results of immune analyses were slightly improved compared to the baseline values in individuals using the probiotics or the pre- and probiotics combination minidrink, however the differences between groups did not reach the significance level. Phagocytosis and killing were clearly and statistically different in individuals that used either placebo or probiotics or pre- and probiotics minidrinks. Therefore, the probiotics and the pre- and probiotics minidrinks have an important effect on innate immunity, resulting in a significant improvement of both phagocytosis and killing. No effect was found on the quality of life of subjects. No special or unusual features of the safety evaluations were found. No serious adverse events were reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living men and women aged 18 to 65 years-old
* History of recurrent herpes labialis at most 3 episodes after exposure to sunlight in the previous 12 months
* Fitzpatrick skin type 1 to 4
* No presence of herpes labialis lesion at the time of recruitment
* Consent to the study and to comply with study product
* Agreement to adhere to the prescribed list of food and nutrients as provided at the start of the study

Exclusion Criteria:

* Presence of acute/terminal disease
* Intolerance for milk protein or lactose
* Daily consumption of probiotic products 1 month before start of the study
* Treatment with acyclovir or other medication believed to interfere with immune responses at the time of the study
* Participation in any herpes UVB reactivation study within the previous three months
* Episode of herpes labialis within 30 days before enrolment in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2009-09-16 (Actual); Study Completion 2009-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence rate of ultraviolet exposure-lesion | Day 42
  Incidence rate of ultraviolet exposure-lesion at at Day 42.

SECONDARY OUTCOMES:
Incidence rate of ultraviolet exposure-lesion | day 35
  Incidence rate of ultraviolet exposure-lesion at at Day 35.
Incidence rate of ultraviolet exposure-lesion | day 49
  Incidence rate of ultraviolet exposure-lesion at at Day 49
Measurement of lesion size (mm2). | Day 35 day 42 Day 49
  Measurement of lesion size as a product of the length and the width of the lesion (measured in mm2) at Day 35 / 42 / 49.
Time to healing (days). | Day 35 day 42 Day 49
  Time to healing defined as either loss of the hard crust or return to normal skin (measured in days) at Day 35 / 42 / 49
Lesion development by classification of lesion stage. | Day 35 day 42 Day 49
  Lesion development by classification of lesion stage. The lesion stages are shown in table 2 of the clinical protocol (adapted from Spruance et al, 2002). In addition, a photo was made at every visit. At Day 35 / 42 / 49
Duration and intensity of pain (10 cm Vas Analogue Scale). | Day 35 day 42 Day 49
  Duration and intensity of pain as recorded by the patient on a visual analogue scale (VAS) of 100 mm, at Day 35 / 42 / 49.
Change in HSV-specific IgG, IgG3, IgG4 and IgE concentrations | Day 49
  HSV-specific IgG1 and IgG3 (Th1) and IgG4 and IgE (Th2) concentrations were analyzed by ELISA at day 49.
Change in HSV-specific CD8+ T cells by pentamers | Day 49
  Immunologic evaluation of HSV-specific CD8+ T cells by pentamers (only on HLA A2-01+ individuals: an estimated 35-40% of individuals fit this criterion) at day 49.
Change in HSV-specific CD8+ T cells by IFN-gamma ELISPOT | day 49
  Immunologic evaluation of HSV-specific CD8+ T cells by IFN-gamma ELISPOT (only on HLA A2-01+ individuals: an estimated 35-40% of individuals fit this criterion) at day 49.
Change in lytic ability of CD8+ T cells | day 49
  Immunologic evaluation of the lytic ability of CD8+ T cells by FACS analyses (perforin, granzymes) (all individuals).
Change in IL-2, IFN-γ, IL10 | day 49
  The following intracellular cytokine concentrations in HSV-stimulated CD4+ cells at day 49:
  * Interleukin-2;
  * Interferon-γ;
  * Interleukin-10.
Change in SF-36 QoL questionnaire. | day 49
  The quality of life was determined by the SF-36 quality of life questionnaire at day 49.
Change in Phagocyte number and activity | day 49
  Phagocyte number and activity as measured by flow cytometry;
Change in NK cell number and activity | day 49
  Natural killer cell number and activity as measured by flow cytometry.